CLINICAL TRIAL: NCT01583439
Title: An Evaluation of the Uptake and Safety of, and Adherence to Antiretroviral Treatment Among Individuals With CD4 ≥ 250 Cells/mm3 and HIV Virus Load ≥ 50,000 cp/mL
Brief Title: The Mochudi Prevention Project ART Protocol
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Accrual.
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Max Essex, Study Principal Investigator, Harvard School of Public Health (HSPH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BHP041; R01AI083036 (NIH)
Record Dates: First submitted 2012-04-11; First posted 2012-04-24 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infections
Keywords: HIV Infections; Acquired Immunodeficiency Syndrome; Anti-HIV Agents; Sexually Transmitted Diseases, Viral; Immunologic Deficiency Syndromes; Immune System Diseases; Anti-Retroviral Agents; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases, Viral; Immunologic Deficiency Syndromes; Immune System Diseases | interventions — Ritonavir; Lamivudine; Zidovudine; efavirenz; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: highly active antiretroviral therapy: Lopinavir/Ritonavir, Lamivudine, Zidovudine, Efavirenz, Tenofovir Disoproxil Fumarate, Emtricitabine — Atripla: one tablet administered orally once daily at bedtime, each tablet comprised of co-formulated: Efavirenz (EFV) 600mg, Emtricitabine (FTC) 200mg, Tenofovir disoproxil fumarate (TDF) 300mg(EFV/FTC/TDF). Note: the study will generally provide the fixed-dose combination Atripla, but it will also be permissible for the same drugs to be used at the same doses as individual components (or as Truvada, coformulated TDF/FTC). Other drug substitutions may be made per the protocol.

SUMMARY:
The goal of the "Mochudi Prevention Project" is to reduce the number of new HIV infections in the village of Mochudi, Botswana by promoting a comprehensive package of interventions that have proven to be effective in preventing the spread of HIV. This antiretroviral treatment (ART) clinical study is nested within the Mochudi Prevention Project, and is being conducted in the north-east segment (NES) of the village of Mochudi. The ART intervention component of the Mochudi Project is designed to determine the uptake of, adherence to, and feasibility of 3-drug combination ART as a component of a package of transmission prevention strategies. The hypotheses are 1) that ART (with 3 antiretrovirals from two classes of drugs) among participants with CD4 ≥ 250 cells/mm3 and VL ≥ 50,000 cp/mL will be acceptable and safe and 2) Eighty percent of eligible participants will agree to start 3-drug ART.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* CD4 cell count ≥ 250 cells/mm3
* HIV-1 RNA ≥ 50,000 cp/mL
* No AIDS-defining illness or other illness that would cause volunteer to be eligible for ART through the Botswana National Program (these volunteers should be referred to the National Program for treatment)
* Age 16 to 64 years
* Botswana citizen
* Resident of the north-east segment of Mochudi
* The following laboratory values obtained within 60 days prior to study enrollment:

  * Absolute neutrophil count (ANC) ≥ 500 cells/mm3.
  * Hemoglobin ≥ 7.0 g/dL.
  * AST (SGOT), ALT (SGPT), and bilirubin ≤ 5 X ULN. Note: if the estimated creatinine clearance (by Cockgroft-Gault equation) is <60 mL/min, then TDF/FTC will be substituted with ZDV/3TC
* Ability to swallow oral medications.
* Ability and willingness of participant to give informed consent (or in case of participants < 18 years of age, ability and willingness to provide assent; and for parent/guardian to provide consent).
* Not currently involuntarily incarcerated.
* Karnofsky performance score ≥ 70 at time of study enrollment.
* If participating in sexual activity that could lead to pregnancy and of reproductive potential, female participants must use two reliable methods of contraception simultaneously, one of which must be a barrier method, while receiving protocol-specified medications, and for 12 weeks after stopping the medications.
* For participants < 18 years of age: Weight of 40kg or more

Exclusion Criteria:

* Receipt at any time prior to study enrollment of > 7 days cumulative treatment with any ARV or combination of ARVs (except ARVs taken for any length of time during pregnancy for the prevention of mother-to-child transmission (pMTCT) or ARVs taken for occupational exposure).
* Current receipt of 3-drug ART for pMTCT
* Allergy/sensitivity to any study drug or its formulations.
* Acute therapy for serious medical illnesses, in the opinion of the site investigator, within 14 days prior to enrollment.

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The proportion of individuals with CD4≥250 cells/mm3 and VL≥50,000 cp/mL who start 3-drug ART
The proportion of patients experiencing Grade 3 or 4 clinical or laboratory adverse events by the end of follow-up
The proportion of participants with excellent adherence (defined as participant self-report of taking at least 95% of doses of antiretrovirals during the previous 4 days, on all assessments) by the end of follow-up

SECONDARY OUTCOMES:
Presence of ARV drug resistance at time of virologic failure on first- and second-line treatment, among participants experiencing virologic failure
Time to first opportunistic infections
Time to death
Time to first episode of non-adherence: the first episode of non-adherence will be the report of the failure of a patient to take 95% of prescribed pills, or participant self-discontinuation of antiretrovirals.
Motivation for / barriers to acceptance of ART will be analyzed descriptively

CONTACTS AND LOCATIONS:
Overall Officials: Max Essex, DVM, PhD, Principal Investigator — Harvard School of Public Health (HSPH); Victor DeGruttola, S.M., Sc.D., Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Deborah Retief Memorial Hospital, Mochudi, Botswana